CLINICAL TRIAL: NCT02896426
Title: Comparison of Collaborative Problem Solving (CPS) and Positive Solutions for Families Groups for Parents of Head Start Preschoolers
Brief Title: Collaborative Problem Solving vs. Positive Solutions for Families in Preschool Parent Groups
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study halted prematurely due to low recruitment and will not resume.
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Caplan Foundation for Early Childhood (Unknown)
Responsible Party: Principal Investigator, Alisha R Pollastri, Director of Research and Evaluation, Think:Kids, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016000948/MGH
Record Dates: First submitted 2016-08-31; First posted 2016-09-12 (Estimated); Last update posted 2018-02-01 (Actual); Status verified 2018-01

CONDITIONS: Child Behavior; Problem Behavior; Family Conflict
Keywords: Parent training; Preschoolers; Behavior problems; Oppositional Defiant Disorder; ODD; Conduct Disorder; CD; Children; Parenting; Collaborative Problem Solving; CPS; Disruptive behavior
MeSH Terms: conditions — Child Behavior; Problem Behavior; Mental Disorders; Oppositional Defiant Disorder; Conduct Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Collaborative Problem Solving (Experimental): Participants will attend parent group sessions led by trained group leaders and learn the Collaborative Problem Solving approach.
  Interventions: Behavioral: Collaborative Problem Solving
- Positive Solutions For Families (Active Comparator): Participants will attend parent group sessions and learn the Positive Solutions for Families approach, a group that is usually offered by Head Start.
  Interventions: Behavioral: Positive Solutions For Families

INTERVENTIONS:
Behavioral: Collaborative Problem Solving — CPS is an approach for understanding and reducing challenging behavior in youth. Under CPS, caregivers are taught to understand and identify the specific neurocognitive skill deficits that underlie their child's challenging behavior. Then the caregivers are taught to interact with the child in a way that solves chronic behavior problems while building the lagging neurocognitive skills to avoid future problems.
  Other Names: CPS
  Arms: Collaborative Problem Solving
Behavioral: Positive Solutions For Families — Positive Solutions for Families groups provide information for families on how to promote children's social and emotional skills, understand their problem behavior, and use positive approaches to help children learn appropriate behavior.
  Arms: Positive Solutions For Families

SUMMARY:
The main objectives of this study are to evaluate the feasibility, acceptability, and effects of a CPS parent group on outcomes for a sample of parents of children ages 3 to 5 compared to outcomes after attending a parenting group that promotes behavioral (operant) parenting. We hypothesize that guardians in the CPS group will report a better understanding of how neurocognitive skills relate to children's behaviors, greater improvements in child functioning and behavior, and greater reductions in parents' stress than those in the comparison group.

DETAILED DESCRIPTION:
Collaborative Problem Solving (CPS) is an evidence-based approach for treating children with behavioral challenges. Unlike traditional models of discipline that use power, control and incentives to facilitate compliance, CPS does not assume that a challenging child lacks motivation for compliance, but instead that the child is motivated to behave well, but simply cannot consistently do so, due to lagging skills in one or more critical neurocognitive domains, such as those related to language and communication skills, attention and working memory skills, emotion- and self-regulation skills, cognitive flexibility skills, and/or social thinking skills. The goal of the intervention is to improve these lagging neurocognitive skills by helping adults and children work toward mutually satisfactory solutions to problems, thereby enhancing flexibility and frustration tolerance in both interaction partners. Any caregiver can use CPS with any child, and CPS can be taught to mental health providers (e.g., therapists, direct care staff), educators (e.g., teachers, administrators), or parents. Common ways to teach CPS to parents include family therapy (one provider teaching one family) or in parent group training (one provider teaching six to ten parents).

Although preschool-aged children have been included in past CPS-related research, they have not been studied separately, and research has not assessed the appropriateness of the current CPS approach for very young children. To address this gap in research, this study will support the development of a parent group curriculum specifically targeting guardians of preschool-aged children, as well as a randomized efficacy trial to evaluate the feasibility, acceptability, and effects of a CPS parent group. Outcome measures from the CPS group will be compared with those from a group that promotes operant behavioral parenting.

Approximately sixty participating guardians will be randomly assigned to attend one of two types of weekly 2-hour groups, each lasting six weeks: either a Collaborative Problem Solving group (N=30; 3 groups) or a Positive Solutions for Families group, a group routinely offered at Head Start programs (N=30; 3 groups). Participants will complete surveys prior to beginning the groups (baseline), upon completion of the group sessions (discharge), and six months after the conclusion of the groups (follow up). Results from these surveys will be compared between groups.

ELIGIBILITY:
Inclusion Criteria:

* Guardian of a child between the ages of three and five currently enrolled at participating Head Start center
* Speaking and writing English at level necessary to complete study requirements

Exclusion Criteria:

* A diagnosis of significant Autism that currently impacts day to day functioning
* A diagnosis of a psychotic disorder including schizophrenia, schizoaffective disorder, schizophreniform disorder
* An intellectual disability that impairs day to day functioning
* Participation in a similar parenting group at the Head Start site within the last year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2016-09; Primary Completion 2017-07-25 (Actual); Study Completion 2017-07-25 (Actual)

PRIMARY OUTCOMES:
Feasibility of a CPS group for parents of preschool-age children | 6 months (immediately after group and 6 months after the group)
  Therapy Attitude Inventory (The TAI is a self-report questionnaire that we will use to measure satisfaction with the parenting groups. We will compare the scores on this measure between the two groups.)

SECONDARY OUTCOMES:
Impact of parenting groups on parenting style | 8 months (changes from baseline, immediately after group, and 6 months after the group)
  Parenting Styles and Dimensions Questionnaire (Measures parenting philosophy and includes scores for authoritative style, authoritarian style, and permissive style.)
Impact of parenting groups on parent emotion regulation | 8 months (changes from baseline, immediately after group, and 6 months after the group)
  Difficulties in Emotion Regulation Scale (Measures emotion regulation skills including nonacceptance of emotional responses, difficulties engaging in goal-directed behaviors, impulse control difficulties, lack of emotional awareness, limited access to emotion regulation strategies, and lack of emotional clarity.)
Impact of parenting groups on the parent child relationship | 8 months (changes from baseline, immediately after group, and 6 months after the group)
  Parent Child Relationship Inventory (Measures how parents view the task of parenting and how they feel about their children. Measures parental support, satisfaction with parenting, communication, limit setting, parent response consistency, and parent social desirability.)
Impact of parenting groups on the parent philosophy | 8 months (changes from baseline, immediately after group, and 6 months after the group)
  Think:Kids Measure of Change Over Time (Measures perceptions of parent-child relationship quality, parenting philosophy, and predictability of youth's challenging behavior.)
Acceptability of a CPS group for parents of preschool-age children | 8 months (changes from baseline, immediately after group, and 6 months after the group)
  Qualitative interviews at each time point
Parent satisfaction with a CPS group for preschool-aged children | 8 months (changes from baseline, immediately after group, and 6 months after the group)
  Qualitative interviews at each time point
Parent satisfaction with a CPS group for preschool-aged children | 8 weeks (immediately after conclusion of group)
  Quantitative parent report of group acceptability at the conclusion of the groups

CONTACTS AND LOCATIONS:
Overall Officials: Alisha R Pollastri, Ph. D., Principal Investigator — Think:Kids at Massachusetts General Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The approach being studied here, Collaborative Problem Solving, is updated and disseminated from Think:Kids at Massachusetts General Hospital. — http://www.thinkkids.org